CLINICAL TRIAL: NCT02272660
Title: Perioperative Parecoxib Administration for Pain Management After Total Knee Arthroplasty and Total Hip Arthroplasty-A Randomized, Placebo-controlled Trial
Brief Title: Parecoxib for Pain Management After Total Knee Arthroplasty and Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Zhihong Wu, Prof, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-503
Record Dates: First submitted 2014-10-17; First posted 2014-10-23 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Pain, Postoperative
Keywords: preemptive analgesia; parecoxib sodium; total knee arthroplasty; total hip arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — parecoxib; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parecoxib sodium (Experimental): The patients in the parecoxib group received a single 40mg dose of parecoxib sodium 30 minutes before incision.
  Interventions: Drug: Parecoxib sodium
- Normal saline injection (Placebo Comparator): The control group received 2 mL normal saline injection at the same time point.
  Interventions: Drug: Normal saline injection

INTERVENTIONS:
Drug: Parecoxib sodium — The patients in the parecoxib group received a single 40mg dose of parecoxib sodium 30 minutes before incision, 9:00 pm on the operation day as well as 9:00 am and 9:00 pm for the next two days after the operation, along with PCIA morphine.
  Other Names: Dynastat
  Arms: Parecoxib sodium
Drug: Normal saline injection — The patients in the control group received 2 mL normal saline injection 30 minutes before Normal saline injection incision, 9:00 pm on the operation day as well as 9:00 am and 9:00 pm for the next two days after the operation, along with PCIA morphine.
  Other Names: Physiological saline
  Arms: Normal saline injection

SUMMARY:
Evaluated the effect of perioperative parecoxib administration on postoperative pain, analgesic use, function recovery, inflammatory response and bleeding risk.

DETAILED DESCRIPTION:
Non-steroid anti-inflammatory drugs are recommended for multimodal postoperative pain management.

We evaluated the effect of perioperative parecoxib administration on postoperative pain, analgesic use, function recovery, inflammatory response and bleeding risk.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients who have underwent primary unilateral total knee arthroplasty (TKA) and total hip arthroplasty (THA).
2. Age between 18-65 years.
3. Chinese ethnicity.

Exclusion Criteria:

1. patients who underwent a reversion or a previous TKA or THA, emergency TKA, or TKA as result of a trauma.
2. patient exhibited allergy to parecoxib sodium.
3. lactating or pregnant.
4. any other conditions not suitable for surgery as evaluated by the surgeon in charge.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the Morphine consumption in each group patients | 4 hours to 6 days after the surgery

SECONDARY OUTCOMES:
To evaluate Patient-Controlled Intravenous Analgesia (PCIA) duration | 4 hours to 6 days after the surgery
To evaluate the Visual Analog Scale (VAS) in each group patients underwent total knee arthroplasty and total hip arthroplasty | 4 hours to 6 days after the surgery
Function recovery of knee Range of Motion (ROM) for patients received surgery | 3 and 6 days after the surgery

OTHER OUTCOMES:
Testing of body temperature,routine blood examination, IL-6 and IL-10 | hospital admission and 1, 3, 6 days after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Wu, Prof, Principal Investigator — PUMC
Locations (1):
- The Peking Union Medical College Hospital, Beijing, Beijing Municipality, China